CLINICAL TRIAL: NCT06593275
Title: Pain Perception in Protection of the Palatal Donor Area After Harvesting a Free Gingival Graft Using Flowable Resin Versus a Self-adhesive Dressing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Especialidades Espiritu Santo (Other)
Responsible Party: Principal Investigator, Antonio Lanata Flores, Assistant Professor, Universidad de Especialidades Espiritu Santo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-ODONT-002B
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Perception of Pain; Protection of the Palate
Keywords: protection of the palate; pain palate; flow resine; self-adhesive dressing

STUDY DESIGN:
Intervention Model Description: The study includes 30 patients who will undergo periodontal or peri-implant surgery with collection of a connective tissue graft from the palate to assess the perceived postoperative pain according to both palatal protection techniques in reference to L. Tavelli et al. 2017. They will be divided into 2 randomized groups, 15 with photocured fluid resin protection and the remaining 15 with a self-adhesive and sutured dressing.
Who Masked: Participant
Masking Description: The patient will not know what protection technique will be used during surgery, but the operator will know at the time prior to surgery with a randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Experimental): This group is defined by the use of a collagen hemostatic sponge and photocured fluid resin for the protection of the palatal donor area by means of an adhesive protocol to the palatal surfaces of the neighboring teeth and fixed with X-suture to improve its stability in the area. A visual analog scale examination will be performed to assess the postoperative pain generated in the palate from day 1 to 14 and ending with the removal of this protection.
  Interventions: Procedure: Protection of the palatal donor area with flowable resin
- Experimental group (Experimental): This group is defined by the use of a collagen hemostatic sponge and a self-adhesive dressing for the protection of the palatal donor area and fixed with an X-shaped suture to improve its stability in the area. A visual analog scale examination will be performed to evaluate the postoperative pain generated in the palate from day 1 to 14 and ending with the removal of this protection.
  Interventions: Procedure: Protection of the palatal donor area with a self-adhesive dressing

INTERVENTIONS:
Procedure: Protection of the palatal donor area with flowable resin — Use of fluid resin for protection of the palatal donor area to assess postoperative pain generated during14 days
  Arms: Control group
Procedure: Protection of the palatal donor area with a self-adhesive dressing — Use of a self-adhesive dressing for protection of the palatal donor area to evaluate postoperative pain generated for 14 days
  Arms: Experimental group

SUMMARY:
The use of a connective tissue graft harvested from the palate is currently one of the most effective and predictable alternatives for the correction of periodontal and peri-implant defects, but the discomfort generated in the palate is sometimes greater than mucogingival surgery. For this reason, we found the need to use different materials for palatal protection. In one group we will use light-cured fluid resin compared to another group a self-adhesive dressing to check which of these materials provides less postoperative pain generated by the harvest of a free gingival graft.

DETAILED DESCRIPTION:
The postoperative pain generated by the harvest of a free gingival graft for the correction of periodontal or peri-implant defects, it's greater when it is not adequately protected and until the reepithelialization of the area is complete. For this reason, it was decided to use two materials to compare the effectiveness in reducing postoperative pain in grafts larger than 15 mm. A control group will be treated with a hemostatic collagen sponge and photocured fluid resin, adhered to the palatal surfaces of the neighboring teeth using an adhesive protocol and X-shaped sutures. Another experimental group will be treated with a hemostatic sponge and placement of a self-adhesive dressing stabilized by X-shaped sutures to ensure its permanence in the mouth. The participants will fill out a daily visual analog scale form for 14 days until the removal of the materials. Finally, the results will be tabulated and compared to provide a conclusion of our study.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients with plaque control less than 20%
* Patients with bleeding on probing less than 10%
* Patients in need of periodontal or peri-implant surgery in the upper or lower jaw
* Not having previous surgeries in the donor area

Exclusion Criteria:

* Pregnant or breastfeeding patients
* Patients with lesions in the palate
* Patients who use prostheses that cover the palate
* Patients with active periodontal disease
* Patients who smoke
* Patients with systemic diseases
* Torus palatinus
* Patients with a history of chemotherapy and radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2029-12-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain perception in the palate | Participants will fill out forms from day 1 after surgery until day 14
  The harvesting of a connective tissue graft from the palate is the gold standard for periodontal and peri-implant surgery, in which the patient reports greater discomfort in this area if it is not properly protected. From this point of view, randomized patients who will receive protection with fluid resin or self-adhesive dressing will be required to fill out a visual analog scale form in which 0 is the minimum pain presented and 10 the maximum pain. The results will be tabulated to make a comparison between both techniques and to verify which one presented the least postoperative pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Especialidades Espiritu Santo, Samborondón, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: No